CLINICAL TRIAL: NCT05724862
Title: Evaluation of Efficacy of Pulpal Anesthesia and Patient Preference Using the Needle-less and Conventional Injection Techniques in Patients With Symptomatic Irreversible Pulpitis in Maxillary Molars: A Randomized Clinical Trial
Brief Title: Efficacy of Pulpal Anesthesia and Patient Preference Using the Needle-less and Conventional Injection Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nader Ramsis, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-11-2022
Record Dates: First submitted 2022-11-25; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Symptomatic Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle-less jet anaesthesia (Experimental): Infiltration anaesthesia without needle
  Interventions: Device: Needle-less jet anaesthesia
- Conventional injection anaesthesia (Active Comparator): Regular infiltration anaesthesia
  Interventions: Device: Conventional Injection Anesthesia

INTERVENTIONS:
Device: Needle-less jet anaesthesia — Infiltration anesthesia without needle depending on injection pressure
  Arms: Needle-less jet anaesthesia
Device: Conventional Injection Anesthesia — Regular Infiltration local anesthesia
  Arms: Conventional injection anaesthesia

SUMMARY:
Pain despite being a physiological experience, is considerably affected by the emotional states, such as anxiety and fear. It was demonstrated that individuals with a high level of anxiety experience difficult anesthesia and more painful procedures during different dental treatments. Besides, the level of anxiety was established as one of the most crucial predictors of dental anesthesia level.

Techniques and equipment such as topical anesthetic, cold spray, applying pressure, vibratory devices, distraction techniques, sedation medications, have been developed and utilized to reduce pain or fear of dental injections or increase the efficacy of anesthesia. However it is the sight and sensation of a needle that was found by almost 25% of patients to be extremely anxiety provoking stimuli in a survey to determine what dental patients truly fear.

Therefore, Needleless devices that were developed to provide anesthesia without injections would reduce patients' apprehension and anxiety levels resulting in a profound anesthesia for a proper duration of time

DETAILED DESCRIPTION:
The aim of the study, treatment procedures, possible side effects and treatment alternatives will be explained to the patients. Patients will be asked to follow the general instructions and sign a printed informed consent. Patients will be asked to fill the outcomes data charts honestly and accurately.

* Eligible patients will be randomly divided into two equal groups according to randomization mechanism: Group 1 (Comfort-In Jet Anesthesia) and Group 2 (Local Infiltration Anesthesia)
* Pre-operative measures (for all groups):

  * Medical and dental history will be obtained from all participants, clinical and radiographic evaluation for each tooth included in this study will be recorded.
  * Clinical diagnosis of symptomatic irreversible pulpitis will be confirmed based on both subjective and objective findings.
  * The operator will explicitly explain the trial steps to the patients, and an informed consent will be signed by patients who accept enrolment.
  * Pain scale chart will be explained to each participant in order to be used after administration of local anaesthesia.
  * Intervention group (G1): Teeth will be anaesthetized using the Comfort-In Jet device by administering 1 ml of 4% Articaine buccally and 0.5 ml palatally.
  * Control group (G2): Teeth will be anaesthetized using conventional infiltration anaesthesia by administering 1 ml of 4% Articaine buccally and 0.5 ml palatally.
  * Each patient will record the level of discomfort during administration of anaesthesia in the pain scale chart (NRS).
  * Profound pulpal anaesthesia will be checked using an electric pulp tester reading every one minute after anesthetic administration up to ten minutes.
  * Teeth that fail to reach profound pulpal anaesthesia will receive a rescue dose of the same anaesthetic solution (4% Articaine) using the conventional injection technique, if needed, intra-ligamentary injection will be used followed by intra-pulpal anaesthesia in case of persistent pain.
  * After confirming profound pulpal anaesthesia single visit root canal treatment will be performed.
  * Access cavity preparation will be done using round burs and tapered diamond stones and patients will be asked to report any pain and/or discomfort during this step. The pain intensity will be recorded on the NRS.
  * Teeth will be isolated with rubber dam and working length will be obtained by an apex locator and confirmed radiographically to be 0.5 to 1 mm from the radiographic apex.
  * All canals will be prepared with crown down techniques using EdgeEndo rotary files depending on the initial size of the canals.
  * Irrigation will be done using 2 ml of 2.5% NaOCl between each two successive files, then, all canals will have a final flush with 5 ml of 17% EDTA for 1 minute followed by 5 ml of distilled water, 5ml of 2.5% NaOCl and finally 5 ml of distilled water in order to remove any residual chemicals from canals.
  * Pain incidence and intensity during mechanical preparation will also be reported by the patients and recorded on the NRS.
  * After complete preparation canals will be dried and obturated in the same visit and teeth will be temporized.
  * Patients will receive postoperative instructions, and will be allowed to call the operator in case of moderate or severe postoperative pain and if needed, an emergency visit will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-50
* Males and females
* Healthy patients whom are categorized as I or II according to The American Society of Anesthesiologists. (ASA I or II)
* Patients accepting to participate in the trial
* Patients who can understand pain scale and can sign the informed consent
* Mature maxillary molars with symptomatic irreversible pulpitis

Exclusion Criteria:

* Medically compromised patients having significant systemic disorders (ASA III or IV).
* Pregnant females
* Teeth with necrotic pulps
* Non-restorable or periodontally hopeless teeth
* Patients on analgesic or anti-inflammatory drugs 12 hours prior to treatment
* Patients allergic to any of the components of the anesthetic solution

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Intra operative pain | Up to One hour
  Using NRS score

SECONDARY OUTCOMES:
Onset of pulpal anaesthesia | Up to Ten minutes
  Electric pulp tester will be used to measure the time taken for gaining profound anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa I Bakry, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No